CLINICAL TRIAL: NCT02602990
Title: Treatment of Cerebral Arteriovenous Malformations With SQUID™ Liquid Embolic Agent
Status: Completed | Type: Observational
Sponsor: Emboflu (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Other Study IDs: SQUID
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Cerebral Arteriovenous Malformations
Keywords: Cerebral; Arteriovenous; Malformation; Embolization; Endovascular
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral AVM treated with SQUID™
  Interventions: Device: SQUID™

INTERVENTIONS:
Device: SQUID™

SUMMARY:
A non-interventional multicentric study for patients with a cerebral AVM for which endovascular treatment is indicated.

DETAILED DESCRIPTION:
This observational study will collect data about the treatment of ruptured, unruptured, untreated or endovascular previously treated AVM's.

Primary endpoint is safety. Safety will be assessed with the number of procedure-related complications occurring during the endovascular treatment until 30 days after the final embolization.

Secondary endpoint is efficacy. Efficacy will be assessed by angiography and clinical outcome assessments (mRS).

For each patient enrolled, data will be collected at inclusion, at each embolization session and at 6 ± 1 months after the end of the endovascular treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must sign the informed consent form prior to the index-procedure. If patient is unable to provide it him- or herself because of the patient's medical condition, the informed consent of the patient's legally authorized representative shall be requested.
2. The patient has an untreated or endovascular previously treated cerebral AVM for which endovascular treatment is indicated.
3. The patient is at least 18 years old.

Exclusion Criteria:

1. Patient is pregnant.
2. Patient with renal insufficiency (GFR < 45 ml/min/1.73 m²)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a cerebral AVM for whom endovascular treatment is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Incidence of complications / adverse events (Safety) | From the start of the procedure until 30 days after procedure
  The safety is assessed with the number of procedure-related complications occurring during endovascular treatment until 30 days after the final embolization session. Procedure-related complications include complications/adverse events related to the procedure or to the device such as but not limited to hemorrhagic and ischemic complications.

SECONDARY OUTCOMES:
Clinical outcome measurement with mRS (Efficacy) | At 6 months after the last treatment session, compared to baseline
  Change of mRS score at 6 months after treatment phase is assessed compared to baseline mRS score.
Degree of targeted portion of AVM occlusion | 6 months
  The degree of the predefined targeted portion of the AVM's occlusion will be assessed angiographically.

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (5):
  - UZ Antwerpen, Edegem
  - Ziekenhuis Oost Limburg (ZOL), Genk
  - AZ Sint-Lucas, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
- Alfried Krupp Krankenhaus, Essen, Germany